CLINICAL TRIAL: NCT06365424
Title: An Open Label Long-Term Study to Evaluate the Safety and Effectiveness of Fenofibrate in Subjects With Primary Biliary Cholangitis (PBC)
Brief Title: Fenofibrate in Patients With Primary Biliary Cholangitis (PBC)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20151230-5-1
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UDCA (Active Comparator)
  Interventions: Drug: UDCA
- UDCA+Fenofibrate (Experimental)
  Interventions: Drug: Fenofibrate; Drug: UDCA

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate (200 mg/day)
  Arms: UDCA+Fenofibrate
Drug: UDCA — Ursodeoxycholic acid (13-15 mg/kg/day)

SUMMARY:
An Open Label Long-Term Study to Evaluate the Safety and Effectiveness of Fenofibrate in Subjects with Primary Biliary Cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent (signed and dated)
* Participated in the PBC study with fenofibrate (NCT02823353)
* Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

* Treatment-related adverse event (AE) leading to fenofibrate discontinuation
* A medical condition, other than PBC, that in the investigator's opinion would preclude full participation in the study or confound its results (e.g., cancer)
* Known history of other liver diseases
* For females, pregnancy or breast-feeding
* Long-term use of immunosuppressive agents
* Any other condition(s) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2017-04-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Through study completion, up to 120 Months
Percentage of patients with biochemical response | Through study completion, up to 120 Months
  The normalisation of Alkaline Phosphatase

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No